CLINICAL TRIAL: NCT03614416
Title: Clinical Trial Testing the BioSerenity Pulse Oximeter (EOXY) Efficacy, Performance and Safety in Healthy Volunteer
Acronym: EOXY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioSerenity (Industry)
Collaborators: NAMSA (Other); Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BIOSERENITY_80601-2-61
Record Dates: First submitted 2018-04-23; First posted 2018-08-03 (Actual); Results first posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-12

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: No randomisation. All subjects will test simultaneously the gold standard and the EOXY device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EOXY device and Gold standard oximter and SaO2 measures (Experimental): Heart rate and SPO2 measures provided from EOXY device Heart rate measures provided from gold standard oximeter. SaO2 measures provided from blood sampling There is only one arm: all subjects have simultaneously three interventions (as required in the European standard ISO 80601-2-61), to qualify a pulse oximeter
  Interventions: Device: EOXY device; Device: Gold standard oximeter; Procedure: SaO2 sampling

INTERVENTIONS:
Device: EOXY device — Sp02 and HR measures from EOXY device are simulateously compared to gold standard measures : Sa02 sampling measures and pulse oximeter gold standard
Device: Gold standard oximeter — Sp02 and HR measures from EOXY device are simulateously compared to gold standard measures : Sa02 sampling measures and pulse oximeter gold standard
Procedure: SaO2 sampling — Sp02 and HR measures from EOXY device are simulateously compared to gold standard measures : Sa02 sampling measures and pulse oximeter gold standard

SUMMARY:
The purpose of the study is to test the performance and safety of the Bioserenity pulse oxymeter EOXY. For that, and in agreement with ISO60601-2-61 norm and FDA regulation, measures of heart rate, with a gold-standard, and SaO2 measures generated by blood samples will be compared with Sp02 and heart rate measures that are generated by our EOXY.

Thirteen healthy subjects will participate in the study in total. Three subjects will be enrolled during a primary phase .They will participate at a secondary phase as well as ten others subjects. The purpose of the primary phase is to test the body area where the measurement can be done. The purpose of the secondary phase is to measure SpO2 and HR in desaturation conditions.

DETAILED DESCRIPTION:
The primary objective is to evaluate and document the SpO2 accuracy of the pulse oximeter equipment, evaluating the performance of the device compared to invasive method blood sampling (SaO2) by CO-Oximeter in healthy subjects during invasive controlled desaturation study at different ranges (100 % to 70% SaO2).

Subject safety during desaturation and saturation period, will be evaluated by reviewing vital sign: heart rate (HR) continuously and blood pressure/temperature between each desaturation plateau.

There are two secondaries objectives, the measurement of the variation of the fraction of inspired oxygen (FiO2), and the validation of the algorithm for data review and analysis.

For the study primary phase, the purpose of this phase is to test the body area where the SpO2 is better detected and define 3 measurement areas. For this, three healthy volunteers will be placed in normal O2 saturation, the SpO2 will be measured using the Bioserenity oximeter (noninvasive method) and will be compared to a gold-standard oximeter CE-marked. The investigator will determine the best area in the body where the SpO2 could be taken for the following subjects.

During a second phase, the measurement of Sp02 and HR with EOXY, will be performed in O2 saturation conditions up to 100% and then in desaturation by plateau from 100 % to 70%. 3 EOXY pulse oximeter recorded the SpO2 at the same time in 3 different areas of the body. As required by the standard, Sp02 measures will be simultaneously compared to SaO2 values measured by blood sampling taken from an indwelling arterial catheter. The HR obtained with EOXY will be compared simultaneously to a gold standard oximeter CE-marked.

As the example in the standard, it was choosen to do the test on the 70-100% range, with 5 plateaus (100%-97%, 97%-92%, 92%-85%, 84%-78%, 77%-70%) and to collect five Sp02 and Sa02 values (blood samples) and five HR measures, per plateau, for each of 13 subjects.

The desaturation will be controlled thanks' the FiO2 measures, that should allow to bring subjects near target levels of desaturation plateau.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject (Man/ Women) > 18 years old
* Subject signed informed consent prior to any screening procedure
* Subject in good health (COHb < 3% , MetHb < 2%, CtHb > 10mg/dL)
* Healthy adult capable of undergoing controlled hypoxemia to the level called for in the protocol with minimal medical risk

Exclusion Criteria:

* Smokers or individuals exposed to high levels of carbon monoxide that result in elevation of carboxy hemoglobin levels
* Individual subject to conditions that result in elevated levels of methemoglobin
* Subject who would be placed at undue medical risk associated with any procedure called for in the protocol
* Subject with open wounds
* Pregnant woman (negative pregnancy test needed)
* Subject allergic to silicon, polyamide and silver yarn
* Subject with cardiorespiratory disorders likely to worsen with thoracic pressure applied by the textile band
* Subject with mental or motor impairment preventing him from expressing pain
* Subject with blood or skin disorder that may impacting results
* Subject with behavioral disorders, too agitated or too aggressive
* Subject with sensorial disorders, insensible to skin pain
* Subject susceptible to tension/pressure based headaches

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: marc FRANCAUX, Principal Investigator — UNIVERSITE CATHOLIQUE DE LOUVAIN
Locations (1):
- Université catholique louvain la neuve, centre sportif, Louvain-la-Neuve, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- EOXY Device and Gold Standard Oximeter and SaO2 Measures: Heart rate and SPO2 measures provided from EOXY device Heart rate measures provided from gold standard oximeter. SaO2 measures provided from blood sampling There is only one arm: all subjects have simultaneously three interventions (as required in the European standard ISO 80601-2-61), to qualify a pulse oximeter
  EOXY device: Sp02 and HR measures from EOXY device are simulateously compared to gold standard measures : Sa02 sampling measures and pulse oximeter gold standard
  Gold standard oximeter: Sp02 and HR measures from EOXY device are simulateously compared to gold standard measures : Sa02 sampling measures and pulse oximeter gold standard
  SaO2 sampling: Sp02 and HR measures from EOXY device are simulateously compared to gold standard measures : Sa02 sampling measures and pulse oximeter gold standard
Period: Overall Study
Arm/Group | EOXY Device and Gold Standard Oximeter and SaO2 Measures
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Healthy subjects (3 patients excluded reducing the number analyzed at 10)
Arm/Group | EOXY Device and Gold Standard Oximeter and SaO2 Measures
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 23.5 [19 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage SPO2 Accuracy Root-Mean Square (ARMS) at Forehead Position
Description: For each desaturation plateau, SpO2 ARMS are calculated by the difference between the investigational pulse oximeter SpO2 measurement and the co-oximeter's SaO2 measurements
Time Frame: 1 day
Population: Subjects respecting the study conditions (no movements, good irrigation) 3 subjects excluded from analysis(no respect of study conditions) so 10 subjects analyzed
Measure: Number; unit: percentage of ARMS (accuracy)
Arm/Group | EOXY Device and Gold Standard Oximeter and SaO2 Measures
Number analyzed (Participants) | 10
percentage of ARMS (accuracy)
  Overall range 70-100% of O2 | 3.91
  97-100% of O2 | 3.08
  97-92% of O2 | 3.36
  92-85% of O2 | 2.85
  84-78% of O2 | 3.48
  77-70% of O2 | 6.21

2. Primary Outcome: Percentage SPO2 Accuracy Root-Mean Square (ARMS) at Torso Position
Description: For each desaturation plateau, SpO2 ARMS (Accuracy Root-Mean Square) are calculated by the difference between the investigational pulse oximeter SpO2 measurement and the co-oximeter's SaO2 measurements
Time Frame: 1 day
Population: as for outcome 1
Measure: Number; unit: percentage of ARMS (accuracy)
Groups:
- EOXY Device and Gold Standard Oximter and SaO2 Measures: SPO2 measures provided from EOXY device SaO2 measures provided from blood sampling There is only one arm: all subjects have simultaneously three interventions (as required in the European standard ISO 80601-2-61), to qualify a pulse oximeter
  EOXY device: Sp02 measures from EOXY device are simulateously compared to gold standard measures : Sa02 sampling measures and pulse oximeter gold standard
  Gold standard oximeter: Sp02 measures from EOXY device are simulateously compared to gold standard measures : Sa02 sampling measures and pulse oximeter gold standard
  SaO2 sampling: Sp02 measures from EOXY device are simulateously compared to gold standard measures : Sa02 sampling measures and pulse oximeter gold standard
Arm/Group | EOXY Device and Gold Standard Oximter and SaO2 Measures
Number analyzed (Participants) | 10
percentage of ARMS (accuracy)
  Overall range 70-100% of O2 | 11.14
  97-100% of O2 | 12.99
  97-92% of O2 | 12.51
  92-85% of O2 | 9.91
  84-78% of O2 | 7.31
  77-70% of O2 | 10.76

3. Primary Outcome: Percentage SPO2 Accuracy Root-Mean Square (ARMS) at BACK Position
Description: as for outcome 1
Time Frame: 1 day
Measure: Number; unit: percentage of ARMS (accuracy)
Groups:
- EOXY Device and Gold Standard Oximeter and SaO2 Measures: SPO2 measures provided from EOXY device SaO2 measures provided from blood sampling There is only one arm: all subjects have simultaneously three interventions (as required in the European standard ISO 80601-2-61), to qualify a pulse oximeter
  EOXY device: Sp02 measures from EOXY device are simulateously compared to gold standard measures : Sa02 sampling measures and pulse oximeter gold standard
  Gold standard oximeter: Sp02 measures from EOXY device are simulateously compared to gold standard measures : Sa02 sampling measures and pulse oximeter gold standard
  SaO2 sampling: Sp02 measures from EOXY device are simulateously compared to gold standard measures : Sa02 sampling measures and pulse oximeter gold standard
Arm/Group | EOXY Device and Gold Standard Oximeter and SaO2 Measures
Number analyzed (Participants) | 10
percentage of ARMS (accuracy)
  Overall range 70-100% of O2 | 6.02
  97-100% of O2 | 7.09
  97-92% of O2 | 6.63
  92-85% of O2 | 6.57
  84-78% of O2 | 5.06
  77-70% of O2 | 3.96

4. Primary Outcome: HR Accuracy Root-Mean Square (ARMS) at Forehead Position
Description: For each desaturation plateau, HR ARMS are calculated by the difference between the investigational pulse oximeter HR measurement and the HR gold standard measurements
Time Frame: 1 day
Population: People respecting study conditions (good irrigation and no movements)
Measure: Number; unit: percentage of ARMS (accuracy)
Arm/Group | EOXY Device and Gold Standard Oximeter and SaO2 Measures
Number analyzed (Participants) | 10
percentage of ARMS (accuracy)
  Overall range 70-100% of O2 | 12.2
  97-100% of O2 | 10.0
  97-92% of O2 | 11.7
  92-85% of O2 | 11.5
  84-78% of O2 | 14.3
  77-70% of O2 | 13.0

5. Primary Outcome: Percentage of HR Accuracy Root-Mean Square (ARMS) at TORSO Position
Description: as for outcome 4
Time Frame: 1 day
Population: People respecting study conditions (good irrigation, no movements)
Measure: Number; unit: percentage of ARMS (accuracy)
Arm/Group | EOXY Device and Gold Standard Oximeter and SaO2 Measures
Number analyzed (Participants) | 10
percentage of ARMS (accuracy)
  Overall range 70-100% of O2 | 32.1
  97-100% of O2 | 30.8
  97-92% of O2 | 31.5
  92-85% of O2 | 31.5
  84-78% of O2 | 30.4
  77-70% of O2 | 36.5

6. Primary Outcome: Percentage of HR Accuracy Root-Mean Square (ARMS) at BACK Position
Description: as for outcome 4
Time Frame: 1 day
Population: People respecting study conditions (good irrigation and no movements)
Measure: Number; unit: percentage of ARMS (accuracy)
Arm/Group | EOXY Device and Gold Standard Oximeter and SaO2 Measures
Number analyzed (Participants) | 10
percentage of ARMS (accuracy)
  Overall range 70-100% of O2 | 21.1
  97-100% of O2 | 22.3
  97-92% of O2 | 24.6
  92-85% of O2 | 19.2
  84-78% of O2 | 19.1
  77-70% of O2 | 20.6

ADVERSE EVENTS:
Time Frame: 2 days for each subject (days of participation)
Arm/Group | EOXY Device and Gold Standard Oximeter and SaO2 Measures
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-05): https://cdn.clinicaltrials.gov/large-docs/16/NCT03614416/Prot_SAP_000.pdf